CLINICAL TRIAL: NCT03424941
Title: TransCatheter Aortic Valve Implantation and Fractional Flow Reserve-Guided Percutaneous Coronary Intervention Versus Conventional Surgical Aortic Valve Replacement and Coronary By-Pass Grafts for Treatment of Patients with Coronary MultiVessel Disease and Aortic Valve Stenosis
Brief Title: The TransCatheter Valve and Vessels Trial
Acronym: TCW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maatschap Cardiologie Zwolle (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9283
Record Dates: First submitted 2018-01-09; First posted 2018-02-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Aortic Stenosis; Multi Vessel Coronary Artery Disease; TAVI; CABG; PCI; Fractional Flow Reserve
Keywords: Aortic Stenosis (AS); Multi Vessel Coronary Artery Disease (MVD); TransCatheter Aortic Valve Implantation (TAVI); Coronary Artery By-pass Grafting (CABG); Percutaneous Coronary Intervention (PCI); Fractional Flow Reserve (FFR); Surgical Aortic Valve Replacement (SAVR)
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FFR-guided PCI and TAVI (Experimental): FFR-guided PCI and subsequently TAVI treatment with the Medtronic CoreValve Evolut R or Medtronic CoreValve Evolut R PRO
  Interventions: Device: FFR-guided PCI and TAVI
- CABG and SAVR (Active Comparator): CABG and SAVR
  Interventions: Device: CABG and SAVR

INTERVENTIONS:
Device: FFR-guided PCI and TAVI — Treatment of subjects with multivessel coronary artery disease and aortic stenosis for FFR-guided PCI and TAVI (Medtronic CoreValve Evolut R or Medtronic CoreValve Evolut R PRO)
  Arms: FFR-guided PCI and TAVI
Device: CABG and SAVR — Treatment of subjects with multivessel coronary artery disease and aortic stenosis for CABG and SAVR
  Arms: CABG and SAVR

SUMMARY:
The trial objective is to investigate whether Fractional Flow Reserve (FFR)-Guided Percutaneous Coronary Intervention (PCI) and TransCatheter Aortic Valve Implantation (TAVI) strategy for treatment of multivessel disease and aortic stenosis will be non-inferior to Coronary Artery By-pass Grafting (CABG) and Surgical Aortic Valve Replacement (SAVR) for a composite primary endpoint of all-cause mortality, stroke, myocardial infarction, coronary or valve re-intervention and life-threatening or disabling bleeding at one year.

DETAILED DESCRIPTION:
Prospective, randomized, controlled, open label, multicenter, international, non-inferiority trial

If the Heart Team decides that a coronary revascularization and aortic valve replacement is needed and the patient complies with inclusion and exclusion criteria then the patient will be randomized in a 1:1 fashion between FFR-guided PCI + TAVI and CABG + SAVR.

Patients will receive optimal medical treatment at discharge. Follow-up will be performed at 30 days and at one year. During the 30 day follow-up visit (after TAVI) patients will be evaluated for symptoms of angina.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic patients aged ≥70 years with aortic stenosis fulfilling one of these criteria (Aortic Valve Area (AVA) ≤1 cm2; mean gradient ≥40 mmHg; Aortic jet velocity >4 m/sec; or Velocity index ≤ 0.25) feasible for treatment by both trans femoral or subclavian approach TAVI as well as conventional SAVR and where the Heart Team decides that treatment is needed (final decision is left to the Heart Team)
2. Presence of ≥2 de novo coronary lesions of ≥50% diameter stenosis on visual estimation located in any of main epicardial coronary arteries, or side branches of a lumen caliber of more than 2 mm or single Left Anterior Descending (LAD) lesion with more than 20 mm length or involving a bifurcation (complex), feasible for treatment with CABG as well as PCI (Heart Team decision)
3. Patients willing and capable to provide written informed consent

Exclusion Criteria:

1. Patients in cardiogenic shock or acute heart failure, requiring inotropic agents during procedure and/or i.v. diuretics <48 hours before procedure
2. Left ventricular ejection fraction <30%
3. Concomitant presence of other than aortic valve disease requiring intervention
4. Previous CABG, SAVR, TAVI or thoracotomy for any other reason
5. Bicuspid or unicuspid aortic valve
6. Recent myocardial infarction (less than 2 weeks)
7. Involvement of left main trifurcation (all three branches being larger than 2 mm)
8. Expected total stent length more 60mm per vessel
9. FFR measurement judged impossible
10. Life expectancy <1 year
11. Known malignancy
12. Contraindication for dual antiplatelet therapy or expected surgical intervention requiring interruption of Dual Antiplatelet Therapy (DAPT) in the first 6 months
13. Reduced renal function (Glomerular Filtration Rate (GFR) <29 ml/min/1.73m2; Kidney Disease Outcomes Quality Initiative (KDOQI) stage 4 and 5)
14. Previous disabling stroke, Transient Ischemic Attack (TIA) in the last 6 months, or known severe stenosis of carotid or vertebral arteries
15. Participation in other investigational clinical trials

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite of all-cause mortality, myocardial infarction, disabling stroke, unscheduled clinically-driven target vessel revascularization, valve re-intervention, and life threatening or disabling bleeding at one year | one year

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE: a composite of cardiovascular mortality, all stroke, myocardial infarction, unscheduled coronary or valve re-intervention) at one year | one year
All-cause mortality and all stroke at 30 days and at one year | 30 days and one year
Life-threatening or disabling bleeding at 30 days and one year | 30 days and one year
Life-threatening or disabling bleeding and major bleeding at 30 days and at one year | 30 days and one year
Rate of conduction disturbances requiring a permanent pacemaker at 30 days and at one year | 30 days and one year
Access-related complications at 30 days | 30 days
Acute kidney injury (Acute Kidney Injury Network (AKIN) classification) at 30 days and at one year | 30 days and one year
Stent thrombosis according to Academic Research Consortium (ARC) criteria (definite and probable) at 30 days and at one year | 30 days and one year
Device success (Valve Academic Research Consortium (VARC) 2 definition) | procedure
Early Safety at 30 days (VARC 2 definition) | 30 days
Early Efficacy at 30 days (VARC 2 definition) | 30 days
Time Related Valve Safety at 30 days (VARC 2 definition) | 30 days
Echocardiographic assessment of prosthetic valve performance at discharge and at one year using the following measures: a) transvalvular mean gradient, b) Effective Orifice Area (EOA), c) degree of prosthetic aortic valve regurgitation | discharge and at one year
Clinically driven revascularisation at 30 days and at one year | 30 days and one year
Change in New York Heart Association (NYHA) class before treatment, at 30 days and at one year | 30 days and one year
Change in Canadian Cardiovascular Society (CCS) class before treatment, at 30 days and at one year | 30 days and one year
Quality of life (Short Form (SF)-36) before treatment and at one year | one year

CONTACTS AND LOCATIONS:
Overall Officials: prof. Elvin Kedhi, MD, PhD, Principal Investigator — Hopital Erasme, Brussels, Belgium
Locations (20):
- Austria (2):
  - Medical University of Graz, Graz
  - General Hospital Vienna, Vienna
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHRU de Lille, Lille
  - Clinique Pasteur, Toulouse
- Universitäres Herz- und Gefäßzentrum UKE Hamburg GmbH, Hamburg, Germany
- Onassis Cardiac Surgery Center, Kallithea, Greece
- Netherlands (6):
  - OLVG, Amsterdam
  - UMCG, Groningen
  - St. Antonius hospital, Nieuwegein
  - Radboudumc, Nijmegen
  - Hagaziekenhuis, The Hague
  - Isala hospital, Zwolle
- Poland (2):
  - Medical University of Silesia, Katowice
  - University hospital Opole, Opole
- Hospital de Santa Cruz, Lisbon, Portugal
- SUSCCH, Banská Bystrica, Slovakia
- Spain (2):
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Clínico Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kedhi E, Hermanides RS, Dambrink JE, Singh SK, Ten Berg JM, van Ginkel D, Hudec M, Amoroso G, Amat-Santos IJ, Andreas M, Campante Teles R, Bonnet G, Van Belle E, Conradi L, van Garsse L, Wojakowski W, Voudris V, Sacha J, Cervinka P, Lipsic E, Somi S, Nombela-Franco L, Postma S, Piayda K, De Luca G, Kolkman E, Malinowski KP, Modine T; TCW study group. TransCatheter aortic valve implantation and fractional flow reserve-guided percutaneous coronary intervention versus conventional surgical aortic valve replacement and coronary bypass grafting for treatment of patients with aortic valve stenosis and complex or multivessel coronary disease (TCW): an international, multicentre, prospective, open-label, non-inferiority, randomised controlled trial. Lancet. 2025 Dec 21;404(10471):2593-2602. doi: 10.1016/S0140-6736(24)02100-7. Epub 2024 Dec 4. PMID 39644913
- [Derived] Kedhi E, Rroku A, Hermanides RS, Dambrink JH, Singh S, Berg JT, van Ginkel DJ, Hudec M, Amoroso G, Amat-Santos IJ, Andreas M, Teles RC, Bonnet G, Van Belle E, Conradi L, van Garsse L, Wojakowski W, Voudris V, Sacha J, Cervinka P, Lipsic E, Somi S, Nombela-Franco L, Postma S, Piayda K, De Luca G, Malinofski K, Modine T. TransCatheter aortic valve implantation and fractional flow reserve-guided percutaneous coronary intervention versus conventional surgical aortic valve replacement and coronary bypass grafting for treatment of patients with aortic valve stenosis and multivessel or advanced coronary disease: The transcatheter valve and vessels trial (TCW trial): Design and rationale. Am Heart J. 2024 Apr;270:86-94. doi: 10.1016/j.ahj.2024.01.010. Epub 2024 Feb 1. PMID 38309610